CLINICAL TRIAL: NCT02313961
Title: Evaluation of Remote Ischemic Conditioning in ST-elevation Myocardial Infarction as Adjuvant to Primary Angioplasty
Brief Title: Remote Ischemic Conditioning in ST-elevation Myocardial Infarction as Adjuvant to Primary Angioplasty
Acronym: RIC-STEMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Braga (Other)
Collaborators: Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HB-CARD-01
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: ST elevation myocardial infarction; Reperfusion injury; Remote ischaemic conditioning
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIC patients (Experimental): Subjects submitted to remote ischaemic conditioning (RIC)
  Interventions: Other: Remote ischaemic conditioning
- No RIC patients (No Intervention): Subjects not submitted to remote ischaemic conditioning (RIC)

INTERVENTIONS:
Other: Remote ischaemic conditioning — Remote ischaemic conditioning is induced by 3 cycles of manual inflation of a blood pressure cuff placed on the left lower limb to 200 mmHg for 5 minutes and then deflation to 0 mmHg for another 5 minutes.
  Arms: RIC patients

SUMMARY:
The primary objective of the RIC-STEMI trial is to assess whether remote ischaemic conditioning (RIC) as an adjunctive therapy during primary percutaneous coronary intervention (PCI) in patients presenting with ST-elevation myocardial infarction (STEMI) can improve clinical outcomes as assessed by death from cardiac-cause or hospitalization for heart failure (HF) for a minimum follow-up period of 12 months.

DETAILED DESCRIPTION:
Ischemic heart disease (IHD) is the leading cause of mortality worldwide, accounting for over 7 million deaths per year. ST-elevation myocardial infarction (STEMI) accounts for nearly one third of acute coronary syndromes. Despite improved STEMI patient care achieved mainly by timely primary percutaneous coronary intervention (PCI) mortality remains unacceptably high, ranging between 6 and 14%. High mortality rates may partly be ascribed to ischemia-reperfusion injury (IRI) which is believed to account for up to 40-50% of infarct size. Several pharmacological alternatives have been attempted to prevent IRI in promising animal experiments nevertheless clinical translation has been disappointing. On the opposite side, ischemic conditioning (IC) by short cycles of ischemia-reperfusion applied before, during or after a major ischemic event has clearly been shown to attenuate IRI in various clinical scenarios. Moreover, even repeated bouts of limb ischemia are cardioprotective, so-called remote IC (RIC). In 2010, Bøtker et al. showed improved myocardial salvage index as assessed by single photon emission computed tomography 30 days after PCI in patients randomly assigned to receive concomitant RIC whereas Rentoukas et al. found higher proportions of ST-segment resolution with adjunctive RIC compared with PCI alone, although significant reductions in troponin I peaks only reached statistical significance in a subgroup undergoing both RIC and morphine therapy combined with PCI. More recently, the group of Bøtker evaluated the long-term effect of RIC on the very same population they initially recruited (166 patients underwent PCI with adjunctive RIC and 167 patients simply underwent PCI) and showed improved long-term prognosis for patients that underwent adjunctive RIC as regards the composite endpoint of adverse cardiac and cerebrovascular events: all-cause mortality, MI, readmission for heart failure (HF), and ischaemic stroke/transient ischaemic attack. However, although very promising, their results are inconclusive as regards cardiovascular mortality and HF development, since the study was not powered to show differences in these clinical events. Large scale studies addressing major adverse cardiovascular events are warranted.

RIC-STEMI is a single-centre, randomized, controlled trial to assess whether RIC as an adjunctive therapy during primary PCI in patients presenting with ST-elevation myocardial infarction (STEMI) can improve clinical outcomes as assessed by death from cardiac-cause or hospitalization for heart failure (HF) for a minimum follow-up period of 12 months.

After enrollment, participants are randomized according to a computer-generated randomization schedule, in a ratio of 1:1 to RIC or no intervention, in blocks of four individuals. RIC is begun at least 10 min before the estimated time of first balloon inflation and its maximum duration is 30 min. Ischemia is induced by 3 cycles of inflation of a blood pressure cuff placed on the left lower limb to 200 mmHg and then deflation to 0 mmHg for another 5 minutes. Apart from temporary moderate pain in the treated thigh, RIC has been shown innocuous.

All patients receive standard of care therapy according to institutional guidelines, namely treatment with 250 mg aspirin intravenously, 600 mg clopidogrel orally and 5000 IU unfractioned heparin intravenously before PCI. The choice of balloons, stent types and PCI procedure as well as the use of glycoprotein IIb/IIIa inhibitors are left to the discretion of the attending physician.

Considering that STEMI is a medical emergency, little time is available. Eligible patients are orally informed and asked to participate in the study. Enrollment will be based on witnessed oral consent and only after the acute phase has been dealt with will a full written informed consent be obtained. Patients are notified at enrollment of their freedom to abandon the study at any time without consequences.

ELIGIBILITY:
Inclusion Criteria:

* STEMI defined as chest pain (or epigastric pain) for more than 30 minutes and either: (i) new ST elevation at the J point in two contiguous leads with the cut-off points of ≥0.2 mV in men or ≥0.15 mV in women in leads V2-V3 or ≥0.1 mV in all other leads, (ii) or new or presumed new left bundle branch block (LBBB)
* Symptom onset not more than 12 h before presentation
* Willingness and capability to provide informed consent

Exclusion Criteria:

* Cardiogenic shock as defined by systemic hypotension (systolic arterial pressure - SAP - below 90 mmHg) and evidence of tissue hypoperfusion
* Post-cardiac arrest status
* Need for mechanical ventilation
* Known peripheral artery disease or evidence of lower limb ischemia
* Recent myocardial infarction (within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2013-03; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Combined outcome of death from cardiac cause or hospitalization for HF on follow-up, including device implantation (implantable cardioverter defibrillator, cardiac resynchronization and left ventricular assist device). | Minimum follow up of 12 months

SECONDARY OUTCOMES:
MI size. | Index hospitalization.
  Estimated by the 48h area under curve of serum troponin I levels
Left ventricular function. | Index hospitalization.
  Assessed by echocardiography within the first 3 days after admission.
Acute kidney injury. | Index hospitalization.
Major adverse cardiovascular events | Minimum follow up of 12 months
  Re-infarction, stroke and revascularisation

CONTACTS AND LOCATIONS:
Overall Officials: António Gaspar, MD, Principal Investigator — Hospital of Braga
Locations (1):
- Hospital of Braga, Braga, Minho, Portugal

REFERENCES:
- [Background] Mandelzweig L, Battler A, Boyko V, Bueno H, Danchin N, Filippatos G, Gitt A, Hasdai D, Hasin Y, Marrugat J, Van de Werf F, Wallentin L, Behar S; Euro Heart Survey Investigators. The second Euro Heart Survey on acute coronary syndromes: Characteristics, treatment, and outcome of patients with ACS in Europe and the Mediterranean Basin in 2004. Eur Heart J. 2006 Oct;27(19):2285-93. doi: 10.1093/eurheartj/ehl196. Epub 2006 Aug 14. PMID 16908490
- [Background] Yellon DM, Hausenloy DJ. Myocardial reperfusion injury. N Engl J Med. 2007 Sep 13;357(11):1121-35. doi: 10.1056/NEJMra071667. No abstract available. PMID 17855673
- [Background] Frohlich GM, Meier P, White SK, Yellon DM, Hausenloy DJ. Myocardial reperfusion injury: looking beyond primary PCI. Eur Heart J. 2013 Jun;34(23):1714-22. doi: 10.1093/eurheartj/eht090. Epub 2013 Mar 27. PMID 23536610
- [Background] Dirksen MT, Laarman GJ, Simoons ML, Duncker DJ. Reperfusion injury in humans: a review of clinical trials on reperfusion injury inhibitory strategies. Cardiovasc Res. 2007 Jun 1;74(3):343-55. doi: 10.1016/j.cardiores.2007.01.014. Epub 2007 Jan 23. PMID 17306241
- [Background] Cheung MM, Kharbanda RK, Konstantinov IE, Shimizu M, Frndova H, Li J, Holtby HM, Cox PN, Smallhorn JF, Van Arsdell GS, Redington AN. Randomized controlled trial of the effects of remote ischemic preconditioning on children undergoing cardiac surgery: first clinical application in humans. J Am Coll Cardiol. 2006 Jun 6;47(11):2277-82. doi: 10.1016/j.jacc.2006.01.066. Epub 2006 May 15. PMID 16750696
- [Background] Hausenloy DJ, Mwamure PK, Venugopal V, Harris J, Barnard M, Grundy E, Ashley E, Vichare S, Di Salvo C, Kolvekar S, Hayward M, Keogh B, MacAllister RJ, Yellon DM. Effect of remote ischaemic preconditioning on myocardial injury in patients undergoing coronary artery bypass graft surgery: a randomised controlled trial. Lancet. 2007 Aug 18;370(9587):575-9. doi: 10.1016/S0140-6736(07)61296-3. PMID 17707752
- [Background] Hoole SP, Heck PM, Sharples L, Khan SN, Duehmke R, Densem CG, Clarke SC, Shapiro LM, Schofield PM, O'Sullivan M, Dutka DP. Cardiac Remote Ischemic Preconditioning in Coronary Stenting (CRISP Stent) Study: a prospective, randomized control trial. Circulation. 2009 Feb 17;119(6):820-7. doi: 10.1161/CIRCULATIONAHA.108.809723. Epub 2009 Feb 2. PMID 19188504
- [Background] Botker HE, Kharbanda R, Schmidt MR, Bottcher M, Kaltoft AK, Terkelsen CJ, Munk K, Andersen NH, Hansen TM, Trautner S, Lassen JF, Christiansen EH, Krusell LR, Kristensen SD, Thuesen L, Nielsen SS, Rehling M, Sorensen HT, Redington AN, Nielsen TT. Remote ischaemic conditioning before hospital admission, as a complement to angioplasty, and effect on myocardial salvage in patients with acute myocardial infarction: a randomised trial. Lancet. 2010 Feb 27;375(9716):727-34. doi: 10.1016/S0140-6736(09)62001-8. PMID 20189026
- [Background] Rentoukas I, Giannopoulos G, Kaoukis A, Kossyvakis C, Raisakis K, Driva M, Panagopoulou V, Tsarouchas K, Vavetsi S, Pyrgakis V, Deftereos S. Cardioprotective role of remote ischemic periconditioning in primary percutaneous coronary intervention: enhancement by opioid action. JACC Cardiovasc Interv. 2010 Jan;3(1):49-55. doi: 10.1016/j.jcin.2009.10.015. PMID 20129568
- [Background] Sloth AD, Schmidt MR, Munk K, Kharbanda RK, Redington AN, Schmidt M, Pedersen L, Sorensen HT, Botker HE; CONDI Investigators. Improved long-term clinical outcomes in patients with ST-elevation myocardial infarction undergoing remote ischaemic conditioning as an adjunct to primary percutaneous coronary intervention. Eur Heart J. 2014 Jan;35(3):168-75. doi: 10.1093/eurheartj/eht369. Epub 2013 Sep 12. PMID 24031025
- [Derived] Gaspar A, Pereira MA, Azevedo P, Lourenco A, Marques J, Leite-Moreira A. Remote ischemic conditioning in ST-elevation myocardial infarction as adjuvant to primary angioplasty (RIC-STEMI): study protocol for a randomized controlled trial. Trials. 2015 Sep 8;16:398. doi: 10.1186/s13063-015-0937-1. PMID 26350480